CLINICAL TRIAL: NCT02864056
Title: A Randomised Controlled Trial Comparing the Effectiveness of Tai Chi Alongside Usual Care With Usual Care Alone on the Postural Balance of Community-dwelling People With Dementia
Brief Title: The TACIT Trial: TAi ChI for People With demenTia
Acronym: TACIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Collaborators: Southern Health NHS Foundation Trust (Other); Dorset HealthCare University NHS Foundation Trust (Other); University of Plymouth (Other); National Institute for Health Research, United Kingdom (Other Government); University of Southampton (Other); Elemental Tai Chi (Unknown); Alzheimer's Society (Other); Solent NHS Trust (Other Government)
Responsible Party: Principal Investigator, Samuel Nyman, Dr Samuel Nyman, Bournemouth University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TACIT001; CDF-2015-08-030 (Other Grant/Funding Number: National Institute for Health Research); 16/WS/0139 (Other: United kingdom Reserach Ethics Committee)
Record Dates: First submitted 2016-08-05; First posted 2016-08-11 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Dementia; Accidental Falls
MeSH Terms: conditions — Dementia | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual care
- Tai Chi (Experimental): Completes 50 hours of Tai Chi, a combination of in-class and at-home practise.
  Interventions: Other: Tai Chi

INTERVENTIONS:
Other: Tai Chi — Ancient Chinese form of mind/body gentle exercise; this will be done while standing to improve postural balance.
  Arms: Tai Chi

SUMMARY:
This is a three-centre parallel group randomised controlled trial with an embedded process evaluation and intervention pilot phase (details not provided in this summary). The overall research question is: Can a Tai Chi exercise programme prevent falls among people with dementia (PWD), specifically among older PWD living at home?

Primary Outcome measure:

• dynamic postural balance (as a surrogate for falls).

Secondary outcome measures:

* to explore the effects of a Tai Chi exercise programme on static and functional postural balance, fear of falling, cognitive functioning, falls, and quality of life. Also to explore the effects of a Tai Chi exercise programme on their informal carer's dynamic and static postural balance, quality of life, and carer burden
* to determine the acceptability and safety of the Tai Chi intervention
* to inform the design of a future definitive clinical trial.

DETAILED DESCRIPTION:
Amongst people aged over 65, people with dementia (PWD) are much more likely to fall, and be injured, than those without dementia. Being injured from falling over is the main reason why older people attend the hospital A&E department. PWD often experience longer hospital stays following a fall, and may become confused which can be stressful for the carer; and a considerable cost to the NHS.

There is evidence that exercise programmes help to prevent falling. Can a Tai Chi exercise programme prevent falls among PWD living at home? We will investigate whether practising Tai Chi over several months improves dynamic postural balance (because it is a good indicator of how likely someone is to fall). People with mild to moderate dementia who live at home are eligible to take part with their regular care-giver as a 'pair'. We will recruit 150 pairs, i.e. 150 people with dementia and their informal caregiver (300 people in total). The PWD must be aged 18 years or older and both must be willing and able to do standing Tai Chi.

At baseline, the researcher will visit the pair at home to assess the participants' balance, memory skills, and general well-being. Pairs will be randomly assigned to either Tai Chi and usual care (intervention) or usual care only (control).

Pairs in the intervention group will practice Tai Chi together in a weekly group class held locally, and at home, and will complete a diary of how much time was spent doing Tai Chi over six months.

All participants will complete diaries showing how often they fell and whether falls caused an injury.

The baseline assessment will be repeated at six months. A researcher will collect feedback from the pair to see whether the intervention could be (further) tailored to the need of PWD and carers. The change in ability to balance over six months will be compared between PWD in each group.

ELIGIBILITY:
Inclusion Criteria:

Person with dementia:

* Aged 18 or above
* Living at home
* Have a diagnosis of a dementia
* Able to do standing Tai Chi (e.g. not be wheelchair bound)
* Willing to attend weekly Tai Chi classes
* Willing to attend a focus group (intervention pilot phase only)

Carer:

* Able to commit to supporting the PWD by participating in data collection throughout the study and in the intervention components if allocated to the intervention group (minimum of 2 times per week in-person, but ideally more)
* Able to do standing Tai Chi (e.g. not be wheelchair bound)
* Willing to attend weekly Tai Chi classes
* Willing to attend a focus group (intervention pilot phase only)

Exclusion Criteria:

Person with dementia

* Living in a care home
* In receipt of palliative care
* Indicate that they have:

  * Severe dementia
  * A Lewy body dementia or dementia with Parkinson's disease
  * Severe sensory impairment
* Are already currently practising (on average once a week or more) or have been practising within the past six months (on average once a week or more) Tai Chi or similar exercise (Qigong, yoga, or Pilates)
* Are currently under the care of or have been referred to a falls clinic for assessment, or are currently attending a balance exercise programme (e.g. Otago classes)
* Lack mental capacity to provide informed consent

Carer:

* Indicate that they have severe sensory impairment
* Lack mental capacity to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go test | 6 months from Baseline

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | 6 months from Baseline
Postural sway | 6 months from Baseline
  Performance while standing on the floor and on a foam mat
Iconographical Falls Efficacy Scale (Icon-Fes, short form) | 6 months from Baseline
  10 item scale of fear of falling
Statue task | 6 months from Baseline
  Visual-spatial cognitive functioning using visual scenes on a small handheld tablet
ICEpop CAPability measure for Older people (ICECAP-O) | 6 months from Baseline
Number and rate of falls | 6 months from Baseline
Number and rate of fallers | 6 months from Baseline
Number and rate of injurious falls | 6 months from Baseline
Zarit Burden Interview (short-form) | 6 months from Baseline
  12 item scale assessing burden on carer
Mini-Addenbrooke's Cognitive Examination (M-ACE) | 6 months from Baseline
  Assess global cognitive functioning

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Nyman, PhD, Principal Investigator — Bournemouth University
Locations (3):
- United Kingdom (3):
  - Memory Assessment Service, Dorset HealthCare University Foundation Trust, Poole, Dorset
  - Solent NHS Trust, Portsmouth, Hampshire
  - Memory Assessment and Research Centre, Southern Health NHS Foundation Trust, Southampton, Hampshire

IPD SHARING:
Plan to Share IPD: Yes
A Data Management Plan will be prepared to facilitate access, sharing and preservation. This will be explicitly referred to in the Statistical Analysis Plan and in the resultant publication of the main trial outcome. This will include specific detail of how potential bona fide research teams will be able to access the following from the CI's institution (Bournemouth University) online repository after an embargo period of approximately 24 months from the publication of the main trial outcome paper.

REFERENCES:
- [Derived] Nyman SR, Casey C, Greenwood N. Hypothesis: Dementia Diminishes Interdependence in Health and Quality of Life Among Spousal Partners. Alzheimer Dis Assoc Disord. 2023 Apr-Jun 01;37(2):174-177. doi: 10.1097/WAD.0000000000000539. Epub 2023 Jan 18. No abstract available. PMID 36706322
- [Derived] Williams J, Nyman S. A secondary analysis of a randomised controlled trial to investigate the effect of Tai Chi on the instrumented timed up and go test in people with mild to moderate dementia. Aging Clin Exp Res. 2021 Aug;33(8):2175-2181. doi: 10.1007/s40520-020-01741-7. Epub 2020 Nov 3. PMID 33141417
- [Derived] Nyman SR, Ingram W, Sanders J, Thomas PW, Thomas S, Vassallo M, Raftery J, Bibi I, Barrado-Martin Y. Randomised Controlled Trial Of The Effect Of Tai Chi On Postural Balance Of People With Dementia. Clin Interv Aging. 2019 Nov 19;14:2017-2029. doi: 10.2147/CIA.S228931. eCollection 2019. PMID 31819385
- [Derived] Nyman SR, Hayward C, Ingram W, Thomas P, Thomas S, Vassallo M, Raftery J, Allen H, Barrado-Martin Y. A randomised controlled trial comparing the effectiveness of tai chi alongside usual care with usual care alone on the postural balance of community-dwelling people with dementia: protocol for the TACIT trial (TAi ChI for people with demenTia). BMC Geriatr. 2018 Nov 3;18(1):263. doi: 10.1186/s12877-018-0935-8. PMID 30390620
- See also: Trial webpage — http://www.bournemouth.ac.uk/tai-chi